CLINICAL TRIAL: NCT06091683
Title: Pilot Study of Adjuvant Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) for the Prevention of Peritoneal Metastases After Curative-intent Surgery for High-risk Colorectal Cancer.
Brief Title: Adjuvant Pressurized Intraperitoneal Aerosol Chemotherapy to Prevent Colorectal Peritoneal Metastases (ProphyPIPAC)
Acronym: ProphyPIPAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 0068/20; 2020-000604-11 (EudraCT Number); BRI D/17/1DB (Other Grant/Funding Number: Fondazione IRCCS Istituto Nazionale Tumori. Milano (Italy)); SC 2020-000604-11_ID_18605 (Other: Agenzia Italiana del Farmaco (AIFA))
Record Dates: First submitted 2023-10-16; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Peritoneal Metastases From Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjuvant pressurized intraperitoneal aerosol chemotherapy (PIPAC) (Experimental): Preliminary laparoscopic exploration of the abdominal cavity and adjuvant pressurized intraperitoneal aerosol chemotherapy (PIPAC) with oxaliplatin and concurrent intravenous infusion of 5-fluorouracil and folinic acid.
  Interventions: Procedure: Pressurized intraperitoneal aerosol chemotherapy (PIPAC)

INTERVENTIONS:
Procedure: Pressurized intraperitoneal aerosol chemotherapy (PIPAC) — Laparoscopic exploration of the abdominal cavity with dissection of adhesions and biopsies of suspect findings (if needed).
  PIPAC will be administered with oxaliplatin (92 mg/m2 body surface area in 150 ml dextrose solution) for 30 minutes under the following spraying conditions: cytostatic application at a rate of 30 ml/min, pressure of 1380 kilo-pascal over 30 minutes, and temperature of 22°C. One hour before the beginning of PIPAC, intravenous infusion of 5-fluorouracil (400 mg/m2) and folinic acid (20mg/m2) will be initiated. Standard protectionist procedures will be adopted to avoid contamination of operators and the environment with nebulized chemotherapy.

SUMMARY:
The objective of this clinical trial is to demonstrate the feasibility and safety of pressurized intraperitoneal aerosol chemotherapy (PIPAC) for the prevention of peritoneal metastases after curative-intent surgery for high-risk colorectal cancer.

DETAILED DESCRIPTION:
This single-arm, single-center, open-label trial enrolls patients after curative-intent surgery for colon adenocarcinoma (proximal to peritoneal reflection), intestinal or mucinous histological type, associated with the following clinical-pathological risk factors for the development of peritoneal metastases: a) stage pT4a, N0-2b, M0 of the Tumor Node Metastasis classification; b) stage pT4b, N0-2b, M0; and c) primary perforated tumor (any T, any N, M0). Eligible patients who will give informed consent undergo laparoscopic pressurized intraperitoneal aerosol chemotherapy (PIPAC) 4 to 8 weeks after primary surgery, followed by adjuvant systemic chemotherapy according to according to current guidelines. After the procedure, patients will be followed-up to assess occurrence of adverse events,survival, peritoneal and systemic disease relapse, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological diagnosis of intestinal type, mucinous or signet ring cell adenocarcinoma of the colon (with upper limit of the tumor above peritoneal reflection);
2. curative (microscopically complete) surgery performed by laparotomy or laparoscopy;
3. presence of at least one of the following risk factors for the development of metachronous peritoneal metastases:

   * perforated primary tumor (any T, N0-2b, M0);
   * primary tumor infiltrating the visceral peritoneum (pT4a, N0-2b, M0), or directly invading adjacent organs (pT4b, N0-2b, M0);
4. age > 18;
5. performance status 2 according to the World Health Organization score;
6. willingness to start adjuvant systemic chemotherapy and post-operative follow-up;
7. Signing of informed consent.

Exclusion Criteria:

1. active sepsis;
2. cardiac function impairment (history of previous heart failure or 40% ejection fraction);
3. renal impairment (serum creatinine >1.5 normal value or creatinine clearance 60 ml/min);
4. liver function impairment (aspartate aminotransferase, alanine aminotransferase, bilirubin > 1.5 normal value);
5. bone marrow function impairment (leukocytes 4000 / mm3, neutrophils 1500 /mm3, platelets 80000/mm3);
6. lung function impairment (diagnosis of severe chronic obstructive pulmonary disease or 50% forced expiratory volume at one second or 40% diffusion capacity of lung for carbon monoxide adjusted for age);
7. extra-abdominal and/or hepatic metastases at the Computed Tomography scan of the chest, abdomen and pelvis with intravenous contrast;
8. severe complications (grade 3-4) after primary cancer surgery;
9. haemorrhagic diathesis or coagulopathy;
10. pregnancy or lactation in progress;
11. psychiatric or neurological conditions such as to preclude protocol procedures; 12) contraindications to laparoscopy; 13) known hypersensitivity to oxaliplatin or other platinum containing compounds and/or to any of their excipients; 14) history of previous malignancies treated in the last three years, excluding cutaneous spinocellular carcinoma and/or basocellular carcinoma; 15) prior pre-operative radio-chemotherapy..

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of adjuvant pressurized intraperitoneal aerosol chemotherapy (PIPAC) | 12 weeks
  The adjuvant PIPAC performed in an early setting after primary surgery will be considered feasible if:
  * the laparoscopic procedure can be completed in 9 patients;
  * the postoperative stay will be three days or shorter in ≥6 patients;
  * the post-operative adjuvant s-CT will begin within 12 weeks of primary surgery in ≥ 9 patients.
Safety of adjuvant pressurized intraperitoneal aerosol chemotherapy (PIPAC) | 30 days
  The adjuvant PIPAC will be considered a well tolerated procedure if:
  * a maximum of one serious treatment-related complication will occur;
  * a maximum of one laparotomy conversion will occur;
  * a maximum of one hospital readmission will occur within 30 days.

SECONDARY OUTCOMES:
Overall survival | 60 months
  Overall survival will be measured from the date of primary surgery to the date of death for any cause or, for patients still alive at the date of the last available follow-up.
Disease-free survival | 60 months
  Disease-free survival will be measured from the date of primary surgery to the date of peritoneal metastasis diagnosis, systemic metastases or death.
Peritoneal disease-free survival | 60 months
  Peritoneal disease-free survival will be measured from the date of primary surgery to the date of peritoneal metastasis diagnosis,

CONTACTS AND LOCATIONS:
Overall Officials: Dario Baratti, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
I confirm that we have a plan to make individual participant data (IPD) available to other researchers through publicly available database
Supporting Information: Study Protocol, CSR
Time Frame: after the completion of the study, for additional 60 months
Access Criteria: upon reasonable request to the principal investigator